CLINICAL TRIAL: NCT04454424
Title: An Open-label Study to Evaluate the Pharmacokinetics, Safety and Tolerability of BAY 1817080 in Participants With Impaired Hepatic Function (Classified as Child-Pugh A, B or C) in Comparison to Matched Controls With Normal Hepatic Function
Brief Title: Study on the Safety of BAY1817080, How it is Tolerated and the Way the Body Absorbs, Distributes and Gets Rid of the Study Drug in Participants With Impaired Liver Function or Normal Liver Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20331
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Endometriosis Related Pain; Overactive Bladder; Diabetic Neuropathic Pain; Refractory or Unexplained Chronic Cough
Keywords: Pharmacokinetics; Safety; Tolerability; Specific population; Subjects with hepatic impairment
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A: Child-Pugh A (Experimental): Participants with mildly impaired hepatic function (Child-Pugh A)
  Interventions: Drug: BAY1817080; Drug: Midazolam
- Arm B: Child-Pugh B (Experimental): Participants with moderately impaired hepatic function (Child-Pugh B)
  Interventions: Drug: BAY1817080; Drug: Midazolam
- Arm C: Child-Pugh C (Experimental): Participants with severely impaired hepatic function (Child-Pugh C)
  Interventions: Drug: BAY1817080; Drug: Midazolam
- Arm D: Normal hepatic (Matched A and B) (Experimental): Participants with normal hepatic function matched to Arm A and B
  Interventions: Drug: BAY1817080; Drug: Midazolam
- Arm E: Normal hepatic (Matched to C) (Experimental): Participants with normal hepatic function matched to Arm C
  Interventions: Drug: BAY1817080; Drug: Midazolam

INTERVENTIONS:
Drug: BAY1817080 — Study intervention BAY1817080 will be administered orally with tablet(s).
Drug: Midazolam — Midazolam will be administered intravenously with dose of 0.1 mg on Day 1.

SUMMARY:
BAY1817080 is currently under clinical development to treat pain related to unexplained chronic cough or chronic cough not affected by a treatment (refractory and/or unexplained chronic cough, RUCC), or a condition where the bladder is unable to hold urine normally (overactive bladder, OAB) or a condition in which tissue similar to the tissue that normally lines the inside of the womb grows outside the womb (endometriosis).

In this study researchers want to learn more about the safety of BAY1817080, how it is tolerated and the way the body absorbs, distributes and gets rid of the study dug given as tablet in participants with mild, moderate or severe hepatic impairment and participants with normal liver function matched for age-, gender-, weight and race.

The study will enroll 36 male and female participants in the age between 18 and 79 years. Participants with mild or moderate hepatic impairment and the matching participants will take multiple oral doses of study drug depending on the study plan. Participants with severe hepatic impairment and the matching participants will take a single oral dose of study drug during the study. Data from this study will provide researcher important information for further development of the study drug in particular on dose recommendation for patients with hepatic impairment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent.
* Participants with a medical history of chronic (For Hepatically Impaired Participants only):

  * documented liver cirrhosis confirmed by histopathology, laparoscopy, fibroscan, CT, MRI or ultrasound, AND
  * hepatic impairment (Child-Pugh A or B or C), AND
  * stable liver disease, i.e. same Child-Pugh class for at least 2 months prior to screening.
* Body mass index (BMI) within the range 18 to 38 kg/m^2 (both inclusive).
* Male or female.
* Women of childbearing potential (WOCBP) must agree to use contraception for the duration of the study. This applies for the time period between signing of the Informed Consent Form until at least 30 days after the last dose of the study drug.
* Capable of giving signed informed consent as described in study protocol which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Any relevant disease (other than those related to hepatic impairment for the hepatic impaired participants) within 4 weeks prior to study drug administration including infections and acute gastro-intestinal diseases (vomiting, diarrhea, constipation) requiring medical treatment.
* Renal failure with an estimated glomerular filtration rate (eGFR) ≤ 35 mL/min, according to Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation.
* Use of strong CYP3A4 and P-glycoprotein inhibitors from 2 weeks before study treatment until last day of blood sampling for pharmacokinetics after study drug administration.
* Use of CYP3A4 and P-glycoprotein inducers from 2 weeks before study treatment until last day of blood sampling for pharmacokinetics after study drug administration.
* Use of drugs which may affect absorption (e.g. loperamide, metoclopramide), and systemic administration of any broad-spectrum antibiotic within 1 week before first study drug administration, unless the drug is part of the mandatory dosing regimen for treatment of hepatic impairment or related conditions.
* Indication or evidence for long QT syndrome; Participants in control arm only: QT interval corrected using Fridericia's method (QTcF) > 450 msec.
* Ascites qualitatively estimated as severe ascites by physical examination, with need of paracentesis; or a recent history of paracentesis.
* Alkaline phosphatase (AP) ≥4 times the upper limit of normal (ULN).
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) in conjunction with gamma-glutamyl transpeptidase (GGT) ≥4 times the ULN (an isolated elevation of GGT above 4 times ULN will not exclude the participant).
* International Normalized Ratio (INR) > 2.7.
* Inability to provide informed consent: Participants with psychiatric disorders, including hepatic encephalopathy >grade 2, e.g. number connection test >80 seconds.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-07-23 (Actual); Primary Completion 2021-06-24 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
AUCu after single dose of BAY1817080 | On day 1
  AUCu: Area under the Curve unbound
Cmax,u after single dose of BAY1817080 | On day 1
  Cmax,u: maximum observed drug concentration in measured matrix after single dose administration (unbound)

SECONDARY OUTCOMES:
Number of subjects with treatment-emergent adverse events | from dosing up to 14 days after end of treatment with study medication
AUC (0-12)md,u after multiple dose of BAY1817080 | From day 6 to day 13
  AUC (0-12)md,u: Area Under the Curve from 0-12 hours at steady state for the multiple dose (unbound)
Cmax,md,u after multiple dose of BAY1817080 | From day 6 to day 13
  Cmax,md,u: Maximum observed drug concentration at steady state for multiple dose (unbound)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/